CLINICAL TRIAL: NCT00518271
Title: A Phase II, Open-Label, Concentration-Controlled, Randomized, 6-Month Study of 'Standard Dose' Tacrolimus + Sirolimus + Corticosteroids Compared to 'Reduced Dose' Tacrolimus + Sirolimus + Corticosteroids in Renal Allograft Recipients
Brief Title: Study Comparing Standard Dose and Reduced Dose Tacrolimus + Sirolimus + Corticosteroids in Renal Allograft Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468E1-100193
Record Dates: First submitted 2007-07-26; First posted 2007-08-20 (Estimated); Last update posted 2007-08-20 (Estimated); Status verified 2007-08

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Sirolimus; Tacrolimus; Adrenal Cortex Hormones

INTERVENTIONS:
Drug: Rapamune® (Sirolimus)
Drug: Tacrolimus
Drug: Corticosteroids — Perioperative

SUMMARY:
This study evaluated renal graft function based on calculated creatinine clearance at 6 months after transplantation in patients receiving a regimen of 'reduced' or 'standard' dose tacrolimus plus sirolimus and corticosteroids.

DETAILED DESCRIPTION:
This study evaluated renal graft function based on calculated creatinine clearance at 6 months after transplantation in patients receiving a regimen of 'reduced' or 'standard' dose tacrolimus plus sirolimus and corticosteroids. Blood serum creatinine, the incidence of biopsy-confirmed acute graft rejection, and patient and graft survival were also evaluated at 6 months post transplantation.

ELIGIBILITY:
Inclusion criteria

* At least 18 years of age
* End-stage renal disease in patients receiving a primary or secondary renal allograft from a cadaveric donor
* Patients with secondary kidney transplant must have maintained their primary graft for at least 6 months

Exclusion criteria

* Planned antibody induction
* Multiple organ transplants
* Patients at high risk of acute rejection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2000-04; Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Graft function as measured by calculated creatinine clearance at month 6 post-transplantation.

SECONDARY OUTCOMES:
Blood serum creatinine, incidence of biopsy-confirmed acute graft rejection, and patient and graft survival at 6 months; presumptive acute rejection; incidence of infection; histologically-confirmed lymphoproliferative disease or malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer